CLINICAL TRIAL: NCT01650272
Title: An Efficacy and Safety Pilot Study Comparing 5% Monoxidil Milky Lotion Versus 5% Minoxidil Solution in Treatment of AGA
Brief Title: Efficacy and Safety Comparing 5% Monoxidil Milky Lotion Versus 5% Minoxidil Solution in Androgenetic Alopecia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Rattapon Thuangtong, Assistant Professor, Siriraj Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SirirajH-006
Record Dates: First submitted 2012-07-23; First posted 2012-07-26 (Estimated); Last update posted 2012-07-26 (Estimated); Status verified 2012-07

CONDITIONS: Objective (Goal); Self-Assessment; Adverse Effects

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5%Minoxidil solution (Experimental): This arm AGA patient receive 5%Minoxidil solution ( Propylene glycol solvent ) to use for 6 month.
  Record efficacy and safety as described.
  Interventions: Drug: 5% Minoxidil solution
- 5%Minoxidil milky lotion (Experimental): This arm AGA patient receive 5%Minoxidil milky lotion to use for 6 month. Record efficacy and safety as described.
  Interventions: Drug: 5% MInoxidil milky lotion

INTERVENTIONS:
Drug: 5% MInoxidil milky lotion — Patient receive 5% MInoxidil milky lotion (Butylene glycol solvent)
  Other Names: MInoxidil milky lotion; MInoxidil milk lotion
  Arms: 5%Minoxidil milky lotion
Drug: 5% Minoxidil solution — Patient receive 5% Minoxidil solution (Propylene glycol solvent )
  Other Names: Minoxidil solution; Minoxidil lotion
  Arms: 5%Minoxidil solution

SUMMARY:
5% Minoxidil lotion was approved for using to stimulate hair growth in male androgenetic alopecia by US FDA science 1988. The mechanism of action still unclear. In general the 5% Minoxidil in solution is the first choice preparation for treatment, therefore allergic contact dermatitis to solution was report up to 5.7% (Ebner H. et al,1995). Propylene glycol which is the main solvent of these solution, was the main responsible to allergic contact dermatitis with positive patch test up to 81.8% (Friedman ES. et al. 2002) One of the alternative solution using butylene glycol as the solvent was invented to solve the problem. In Siriraj hospital the investigators using this new solvent and made our in house product called 5% Minoxidil milky lotion. However the efficacy and safety of the new solution have not been investigated. This study is conducted to evaluated efficacy and safety of 5% Minoxidil milky lotion compare with the classic solution in male androgenetic alopecia.

DETAILED DESCRIPTION:
The 5% Minoxidil in solution is the first choice preparation for treatment for Androgenetic Alopecia (AGA), 5% Minoxidil milky lotion is the alternative solution using butylene glycol as the solvent to solve allergic contact dermatitis problem. In Siriraj hospital the investigators using this new solvent and made our in house product called he efficacy and safety of the new solution have not been investigated. This study is conducted to evaluated efficacy and safety of 5% Minoxidil milky lotion compare with the classic solution in male androgenetic alopecia.

ELIGIBILITY:
Inclusion Criteria:

* New case male AGA
* Classification Norwood III vertex or IV

Exclusion Criteria:

* Have previous AGA treatment in 6 month prior
* Complicated case with other disease condition effect hair such as Anemia, DM, Chronic alcoholism, Autoimmune disease, Thyroid disease, previous GI surgery etc.
* Other scalp lesion such as Psoriasis, Tinea capsitis
* Psychological disorder including trichotillomania

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-02 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy of 5%Minoxidil milky lotion compare to 5%Minoxidil solution | 6 month
  1. Target area hair evaluation
     * Hair density (Digital image, DinoLite pro)
     * Hair diameter (Electronic outside micrometer)
     * Hair count vellus/ non-vellus ratio
  2. Global photographic review (by 2 Experienced Dermatologist)
  3. Patient self evaluation ( 7point scale )

SECONDARY OUTCOMES:
Side effect of topical minoxidil | 6 month
  Record side effect such as Erythema, Dryness, Pruritus, Scaling, etc.

OTHER OUTCOMES:
Weight of topical minoxidil milky lotion / minoxidil lotion | 6 month
  Measure weight of topical minoxidil milky lotion / minoxidil lotion to confirm using of patient

CONTACTS AND LOCATIONS:
Overall Officials: Rattapon Thuangtong, MD, Principal Investigator — Department of Dermatology, Faculty of Medicine Siriraj Hospital, Mahidol University
Locations (1):
- Siriraj Hospital, Bangkok, Bangkok, Thailand